CLINICAL TRIAL: NCT01867242
Title: PROJECT 4: CLINICAL TRIAL METHODS FOR ASSESSING A TOBACCO PRODUCT Part of "MODELS FOR TOBACCO PRODUCT EVALUATION
Brief Title: Methods Project 4: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012NTLS050; 5U19CA157345 (NIH)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2023-04-25 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Smoker
Keywords: cigarette; snus; smoking; tobacco
MeSH Terms: conditions — Smoking | interventions — Tobacco Products; Tobacco, Smokeless

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Brand Cigarette (Experimental): Smoking usual brand cigarette controls, who after 8-weeks will be offered Camel Snus and instructed for partial or complete substitution of cigarettes (subject's choice);
  Interventions: Other: Cigarettes
- Complete Substitution (Experimental): Use snus in place of cigarettes
  Interventions: Other: Snus
- Partial Substitution (Snus and Cigarettes) (Experimental): Use snus and cigarettes how ever you like
  Interventions: Other: Cigarettes; Other: Snus

INTERVENTIONS:
Other: Cigarettes — Smoke their usual brand of cigarettes and follow their normal patterns of use.
  Arms: Partial Substitution (Snus and Cigarettes); Usual Brand Cigarette
Other: Snus — Winterchill or Robust flavors
  Other Names: Camel Snus
  Arms: Complete Substitution; Partial Substitution (Snus and Cigarettes)

SUMMARY:
Cigarette smokers who are eligible will enter a Camel Snus sampling phase. Smokers interested in continuing with the study after the sampling phase will undergo a 2 week baseline assessment phase and will then be randomized to one of the three experimental conditions for 8 weeks. Tobacco use patterns, subjective responses to product, and nicotine and toxicant exposure will be assessed.

DETAILED DESCRIPTION:
Baseline smoking period: Subjects will be required to attend 2 baseline clinic visits where baseline assessments will be captured including a record of their cigarette or other tobacco intake on a daily basis using an interactive voice response system (IVR).

Experimental Period: After the baseline assessment, subjects will be randomized to one of five experimental conditions: 1) smoking usual brand cigarette controls, who after 8-weeks will be offered Camel Snus to use as they will for 8 more weeks; 2) complete substitution (i.e., no smoking) and use snus instead ; 3) partial substitution - use of both snus and cigarettes as you like. Snus, but not cigarettes, will be provided to subjects at the clinic visits. Subjects will attend clinic visits over the next 8 weeks where tobacco use patterns and biomarker data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are at least 18 years of age;
* Daily smoker;
* Generally good health;
* Subject has provided written informed consent to participate in the study (adolescents under the age of 18 will be excluded because this project involves continued use of tobacco products and new tobacco products);

Exclusion Criteria:

* Unstable health
* Pregnant or breastfeeding (due to toxic effects from tobacco products).
* Unable to read for comprehension or completion of study documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (3):
- United States (3):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Roswell Park Cancer Center, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Smokers were recruited from Minneapolis, Minnesota; Columbus and Coshocton, Ohio, and Buffalo, New York between May 2013 and August 2016. Internet and local media advertisements read: "Smokers who want to try a new oral tobacco product are needed for a research study that may reduce their exposure to harmful tobacco smoke."
Pre-assignment Details: After 1 week, participants returned to the clinic with snus tins and unused snus pouches. Tobacco use over the past week was assessed and participants completed self-report questionnaires. Participants who used at least seven snus pouches (based on potential use of one pouch per day) and continued to smoke were eligible to enter the clinical trial. These criteria were withheld from participants to ensure an unbiased willingness to use snus.
Period: Overall Study
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
Started | 64 | 60 | 26
Completed | 40 | 44 | 18
Not Completed | 24 | 16 | 8
Not completed — Lost to follow-up, personal reasons | 24 | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette | Total
Number analyzed (Participants) | 64 | 60 | 26 | 150
Age, Continuous [Mean (Full Range); unit: years] | 42.5 [18 to 83] | 42.0 [18 to 64] | 47.0 [23 to 68] | 43.5 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 13 | 65
  Male | 36 | 36 | 13 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 16 | 11 | 43
  White | 44 | 43 | 15 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 64 | 60 | 26 | 150
Mean cigarettes per day (CPD) [Mean (Full Range); unit: Cigarettes Per Day] | 14.0 [4.3 to 34.4] | 11.7 [6.0 to 39.9] | 12.1 [5.6 to 31.5] | 12.3 [4.3 to 39.9]
Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Full Range); unit: units on a scale] — The FTND is a self-report measure of nicotine dependency. Scores range from 0-8 with higher scores indicating more dependency.
  units on a scale | 3.0 [2 to 6] | 3.0 [0 to 7] | 3.0 [1 to 6] | 3.0 [0 to 7]
Total Nicotine Equivalents (TNE) [Median (Full Range); unit: nmol/mg] | 58.3 [18.5 to 383.1] | 55.9 [0.04 to 307.3] | 65.7 [5.4 to 152.4] | 59.1 [0.04 to 383.1]

OUTCOME MEASURES:

1. Primary Outcome: Smoke-free Days
Description: Number of days subjects smoked no cigarettes during the intervention was compared between groups.
Time Frame: 8 weeks (56 (+/-5) days)
Measure: Median (Full Range); unit: days
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
Number analyzed (Participants) | 64 | 60 | 26
days | 14.5 [0 to 61] | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: CEMA (2-cyanoethylmercapturic Acid)
Description: 2-cyanoethylmercapturic acid (CEMA) is a biomarker for exposure to acrylonitrile, a volatile organic compound, and is sensitive to changes in cigarette smoke exposure.
Time Frame: 8 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mg per creatinine
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
Number analyzed (Participants) | 24 | 38 | 15
pmol/mg per creatinine | 248.1 [142.7 to 431.2] | 438.8 [365.0 to 657.5] | 594.6 [441.9 to 800.0]

3. Secondary Outcome: Total Nicotine Exposure
Description: Urinary total nicotine equivalents, the molar sum of nicotine and six metabolites, accounts for more than 90% of a nicotine dose
Time Frame: 8 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/mg
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
Number analyzed (Participants) | 24 | 39 | 16
nmol/mg | 46.7 [32.5 to 67.0] | 65.0 [53.1 to 79.4] | 63.4 [42.7 to 94.0]

4. Secondary Outcome: Urinary Total NNAL
Description: Urinary 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol and its glucuronides (total NNAL) is a metabolite of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), one of the group of chemicals termed tobacco-specific N-nitrosamines (TSNA)
Time Frame: 8 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mg creatinine
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
Number analyzed (Participants) | 24 | 39 | 16
pmol/mg creatinine | 1.43 [1.07 to 1.91] | 1.27 [1.01 to 1.61] | 1.38 [0.91 to 2.08]

ADVERSE EVENTS:
Time Frame: Adverse events related to study product reported over 8 weeks of snus product use.
Groups:
- Complete Substitution: Substitute snus in place of all cigarettes
  Snus: Winterchill or Robust flavors
- Partial Substitution (Snus and Cigarettes): Substitute snus for cigarettes ad libitum
  Cigarettes: Smoke their usual brand of cigarettes and follow their normal patterns of use.
  Snus: Winterchill or Robust flavors
- Usual Brand Cigarette: Smoking usual brand cigarette controls
  Cigarettes: Smoke their usual brand of cigarettes and follow their normal patterns of use.
Arm/Group | Complete Substitution | Partial Substitution (Snus and Cigarettes) | Usual Brand Cigarette
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/60 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/64 | 0/60 | 0/26
Other Adverse Events (participants affected / at risk) | 5/64 | 1/60 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete Substitution (N=64) | Partial Substitution (Snus and Cigarettes) (N=60) | Usual Brand Cigarette (N=26)
Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | NA (0) | NA (0) — Auto accident unrelated to study product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete Substitution (N=64) | Partial Substitution (Snus and Cigarettes) (N=60) | Usual Brand Cigarette (N=26)
Hearburn/reflux (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Gum sensitivity (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT01867242/Prot_SAP_000.pdf
  • Informed Consent Form (2013-10-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT01867242/ICF_001.pdf